CLINICAL TRIAL: NCT00629967
Title: A Randomized, Open Labeled, Active-Controlled Trial of 24-Week Versus 48-Week Courses of Peg-Interferon Alpha Plus Ribavirin for Genotype-1 Infected Chronic Hepatitis C Patients
Brief Title: A Randomized Trial of 24-Week Versus 48-Week Courses of Peginterferon Plus Ribavirin for HCV Genotype-1 Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: MING-LUNG YU, Kaohsiung Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUH-IRB-94045
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-01

CONDITIONS: Chronic Hepatitis C; Genotype
Keywords: chronic hepatitis C; genotype 1; rapid virological response; sustained virological response; peginterferon; ribavirin; treatment duration
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Eligible patients will be randomized into two groups with a ratio of 1:1 (Arm A & B)
  Interventions: Drug: pegylated interferon alpha 2a and ribavirin
- B (Active Comparator): Eligible patients will be randomized into two groups with a ratio of 1:1 (Arm A & B)
  Interventions: Drug: Pegylated interferon alfa-2a and ribavirin

INTERVENTIONS:
Drug: pegylated interferon alpha 2a and ribavirin — pegylated interferon alpha 2a 180 mcg/week and ribavirin 1000-1200 mg/day for 48 weeks
  Other Names: PEGASYS®
  Arms: A
Drug: Pegylated interferon alfa-2a and ribavirin — Pegylated interferon alfa-2a 180 mcg/week and Ribavirin 1000-1200 mg/day for 24 weeks, follow up for 24 weeks
  Other Names: PEGASYS®
  Arms: B

SUMMARY:
The purposes of this study are:

1. To evaluate whether treatment with peginterferon and ribavirin for 24 weeks is sufficient to achieve a sustained virological response (SVR) rate comparable to that observed with the standard treatment duration of 48 weeks, in hepatitis C virus genotype 1 (HCV-1) patients achieving a rapid virologic response (RVR; <50 IU/mL HCV RNA at week 4) at 4 weeks.
2. To investigate the role of on-treatment virological responses among patients with 24 or 48 weeks treatment.

DETAILED DESCRIPTION:
Peginterferon and ribavirin combination treatment has been recommended for all patients infected with HCV, but the treatment duration varies depending on the HCV genotype. Recommended treatment for patients with HCV-1 infection is pegylated interferon plus ribavirin for 48 weeks and 24 weeks for HCV-2/3. A RVR is a strong predictor of SVR. Previous studies have demonstrated that for HCV-2/3 patients who had a RVR, a shorter duration of treatment with peginterferon plus standard dose of ribavirin over 14 weeks is as effective as a 24-week treatment regimen. These findings have questioned whether shorter treatment duration can yield high SVR rates for HCV-1 pts with an RVR.

The primary aim of the present study is to evaluate whether treatment with peginterferon and ribavirin for 24 weeks is sufficient to achieve an SVR rate comparable to that observed with the standard treatment duration of 48 weeks, in HCV-1 patients achieving an RVR at 4 weeks.

The secondary aim is to investigate the role of on-treatment virologic responses among patients with 24 or 48 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, 18-65 years of age
* Patients have never been treated with traditional interferon plus ribavirin or peginterferon plus ribavirin
* Serologic evidence of chronic hepatitis C infection by an anti-HCV antibody test
* Detectable serum HCV-RNA and HCV viral genotype 1
* Liver biopsy findings consistent with the diagnosis of chronic hepatitis C infection with or without compensated cirrhosis (Exception: hemophiliacs in whom biopsy is medically contra-indicated do not require biopsy.)
* Elevated serum alanine transaminase (ALT) levels for at least two measurements within 6 months preceding the trial entry.
* Compensated liver disease (Child-Pugh Grade A clinical classification)
* Neutrophil count >1500/mm3, platelet count >9×104/mm3, hemoglobin level >12 g/dL for men and >11 g/dL for women, serum creatinine level <1.5 mg/dL
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug
* All fertile males and females receiving ribavirin must be using two forms of effective contraception during treatment and during the 6 months after treatment end

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* Therapy with any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) 6 months prior to the first dose of study drug
* Any investigational drug 6 weeks prior to the first dose of study drug
* Co-infection with active hepatitis A, hepatitis B and/or human immunodeficiency virus (HIV)
* History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* Signs or symptoms of hepatocellular carcinoma
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* Neutrophil count <1500 cells/mm3 or platelet count <90,000 cells/mm3, Hgb <11 g/dL in women or <12 g/dL in men at screening
* Any patient with major thalassemia
* Serum creatinine level >1.5 times the upper limit of normal at screening
* History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease, chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* History of thyroid disease poorly controlled on prescribed medications, elevated thyroid stimulating hormone (TSH) concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease
* Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration)
* Evidence of drug abuse (including excessive alcohol consumption) within one year of study entry
* Inability or unwillingness to provide informed consent or abide by the requirements of the study
* Male partners of women who are pregnant
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4 g/dL (as may be seen with ribavirin therapy) would not be well-tolerated
* Patients with HCV genotype other than 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Efficacy - Sustained virological response (SVR), HCV RNA seronegative by PCR throughout 24-week off-treatment period. | 2 years

SECONDARY OUTCOMES:
Safety - adverse event rate and profile | 2 years
Early virological response (EVR), by PCR-negative or 2 logs decline from baseline at week 12 | 2 years
Rapid virologic response (RVR), HCV RNA seronegative by PCR at week 4. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lung Yu, MD, PhD, Principal Investigator — Kaohsiung Medical University; Chia-Yen Dai, MD, Ms, Principal Investigator — Kaohsiung Municipal Hsiao-Kang Hospital; Chang-Fu Chiu, MD, Principal Investigator — Paochien Hospital; Jee-Fu Huang, MD, Principal Investigator — Foo Yin Hospital
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Dalgard O, Bjoro K, Hellum KB, Myrvang B, Ritland S, Skaug K, Raknerud N, Bell H. Treatment with pegylated interferon and ribavarin in HCV infection with genotype 2 or 3 for 14 weeks: a pilot study. Hepatology. 2004 Dec;40(6):1260-5. doi: 10.1002/hep.20467. PMID 15558712
- [Background] Strader DB, Wright T, Thomas DL, Seeff LB; American Association for the Study of Liver Diseases. Diagnosis, management, and treatment of hepatitis C. Hepatology. 2004 Apr;39(4):1147-71. doi: 10.1002/hep.20119. No abstract available. PMID 15057920
- [Background] Hadziyannis SJ, Sette H Jr, Morgan TR, Balan V, Diago M, Marcellin P, Ramadori G, Bodenheimer H Jr, Bernstein D, Rizzetto M, Zeuzem S, Pockros PJ, Lin A, Ackrill AM; PEGASYS International Study Group. Peginterferon-alpha2a and ribavirin combination therapy in chronic hepatitis C: a randomized study of treatment duration and ribavirin dose. Ann Intern Med. 2004 Mar 2;140(5):346-55. doi: 10.7326/0003-4819-140-5-200403020-00010. PMID 14996676
- [Background] Fried MW, Shiffman ML, Reddy KR, Smith C, Marinos G, Goncales FL Jr, Haussinger D, Diago M, Carosi G, Dhumeaux D, Craxi A, Lin A, Hoffman J, Yu J. Peginterferon alfa-2a plus ribavirin for chronic hepatitis C virus infection. N Engl J Med. 2002 Sep 26;347(13):975-82. doi: 10.1056/NEJMoa020047. PMID 12324553
- [Derived] Yu ML, Dai CY, Huang JF, Chiu CF, Yang YH, Hou NJ, Lee LP, Hsieh MY, Lin ZY, Chen SC, Hsieh MY, Wang LY, Chang WY, Chuang WL. Rapid virological response and treatment duration for chronic hepatitis C genotype 1 patients: a randomized trial. Hepatology. 2008 Jun;47(6):1884-93. doi: 10.1002/hep.22319. PMID 18508296